CLINICAL TRIAL: NCT01423630
Title: Supplementation of Probiotics and Fruit Fibre to Patients With Fatty Liver
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible patients and study staff
Sponsor: Region Skane (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008/517
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Fatty Liver
Keywords: fatty liver; probiotics; Lactobacillus; fruit; fibre; dietary intervention; obesity
MeSH Terms: conditions — Fatty Liver; Obesity | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotics and fruit fibre (Experimental): Probiotics and fruit fibre
  Interventions: Dietary Supplement: Probiotics and fruit fibre

INTERVENTIONS:
Dietary Supplement: Probiotics and fruit fibre — probiotics and fruit fibre

SUMMARY:
Probiotics and fruit fibre are given for 12 weeks to patients with fatty liver disease.

The hypothesis is that probiotic bacteria and fruit fibre affect the gut microbial composition in a positive manner. The improved ecological system is believed to contribute to improved liver health and thereby counteract fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* be able to participate in magnetic resonance imaging

Exclusion Criteria:

* unable to understand oral and written information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Improved and normalized liver status | after 12 weeks intervention
  normalized concentrations of liver enzymes in plasma. Magnetic resonanse imaging (compared to magnetic resonanse imaging before intervention) will also be used in the investigation of improved liver status.

SECONDARY OUTCOMES:
Changes in the gut bacterial flora | after 12 weeks intervention
  Changes and differences of the gut bacterial flora will be addressed in detail, e.g. changes in concentration of specific bacterial groups (e.g. Lactobacillus) before and after the intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Malmo, Sweden